CLINICAL TRIAL: NCT03401437
Title: Quality of Life Assessment of Women Undergoing Laparoscopic Removal of Essure System : a Before-and-after Study
Brief Title: Quality of Life Assessment Before and After Essure Removal
Acronym: ESSURE
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: La Conception Hospital - Marseille - France (Unknown); Public Assistance - Marseille Hospitals (Unknown); Aix Marseille Université (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0154
Record Dates: First submitted 2017-09-26; First posted 2018-01-17 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Patients Presenting Essure Device Attributed Symptoms
Keywords: adverse effects; Salpingectomy; Essure® device ablation; Cornual resection
MeSH Terms: interventions — 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohorte: Patients seen in consultation between January 2017 and August 2017, who have already completed the SF-36 questionnaire (pre-operative, M1 and M3), the HAD and ANSM questionnaires (pre-operative and M3)
- Prospective cohorte: Patients seen in consultation between August 2017
  Interventions: Behavioral: SF-36; Behavioral: HAD; Other: ANSM

INTERVENTIONS:
Behavioral: SF-36 — Evaluation of the quality of life with an auto-questionnaire validated, with 8 dimensions: physical activity ; limitations due to physical condition; physical pain; perceived health; vitality; life and relationship with others; limitations due to physical condition; psychic health as well as the assessment of perceived health compared to a year ago. Evaluation done pre-operatively, at M1 and M3
  Other Names: Short Form 36 Health Survey questionnaire
  Groups: Prospective cohorte
Behavioral: HAD — Evaluation of anxiety and depression with a scale validated with 14 items assess between 0 and 3. Evaluation done pre-operatively and at M3.
  Other Names: Hospital Anxiety and Depression scale
  Groups: Prospective cohorte
Other: ANSM — Additional information requested by the ANSM (french National Agency for Medicines and Health Products Safety) following a materiovigilance report. Evaluation done pre-operatively and at M3.
  Other Names: ANSM questionnaire
  Groups: Prospective cohorte

SUMMARY:
To evaluate quality of life before and after laparoscopic removal of the Essure® system. Women who complain about symptoms attributed to the Essure® device are expected to have an improved quality of life postoperatively.

DETAILED DESCRIPTION:
Tubal sterilization is a widely used method of contraception. The hysteroscopic sterilization method (Essure®; Bayer, Germany) was approved in 2007 in France. Increasing patients reports of complications, such as bleeding pain, allergies, fatigue or articular pain have raised concerns about the safety device. Women suffering of alleged complications of the Essure® device ask for surgical removal. But, only few studies have assessed Essure® removal in terms of quality of life. This observational study contains two parts will be conducted at two academic tertiary care center (Montpellier - Marseille):

* a prospective part having received a favorable opinion from a Committee for the Protection of Persons,
* and a retrospective part having received a favorable opinion from the Institutional Review Board (IRB), local ethics committee

Patients: Women requesting surgical management for removal of Essure® for alleged adverse effects.

Assessment tools :

Quality of life with the Short Form 36 (SF-36) Health Survey questionnaire (pre-operatively and at 1 and 3 months) Hospital Anxiety and Depression (HAD) scale (pre-operatively and 3 months)

Preoperative imaging, procedure characteristics, including the Essure® removal method, operative findings, perioperative complications, histopathologic report, and length of hospital stay will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients carrying Essure®
* Patients requesting surgical removal of Essure®
* Patients with adverse effect
* Being affiliated or benefiting from a French social security system

Exclusion Criteria:

- Patients with guardianship or curators

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with definitive sterilization by Essure®
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-11-16 (Actual)

PRIMARY OUTCOMES:
Improving the quality of life between pre and post-operative at 3 months | 3 months after the surgery
  The quality of life is measure with Short Form (36) Health Survey Questionnaire

SECONDARY OUTCOMES:
General disorders and anxiety or depression | One month before surgery and 3 months after surgery.
  General disorders and anxiety or depression (by questionnaire HAD)
Performance of 3D ultrasound | Preoperatively
  Estimate the performance of preoperative 3D ultrasound to identify a poor implantation of the Essure® found in Preoperatively
Allergy to components | Before removing the sterilization devices (Essure®)
  Reaction to metals: Estimate the prevalence of contact allergy to components through skin tests
Allergy to components | During surgical removal
  Reaction to metals: to estimate the prevalence of Nickel release by the Essure® , by the analysis of the surgical parts
Defects in installation or secondary migration | during surgery
  Estimate the prevalence of Essure® deposition or secondary migration defects

CONTACTS AND LOCATIONS:
Overall Officials: PATRICE PC CROCHET, PhD, Study Director — University Hospital, Montpellier
Locations (2):
- France (2):
  - Public Assistance - Marseille Hospitals, Marseille
  - Montpellier University Hospital, Montpellier